CLINICAL TRIAL: NCT00264901
Title: Impact of a Self-Adjusted Titration Guideline in Subjects With Type 2 Diabetes Mellitus: A Treat-to-Target of the Efficacy and Safety of Levemir® (Insulin Detemir [rDNA Origin] Injection) (PREDICTIVE™ 303)
Brief Title: Comparison of Self Adjustment Versus Standard of Care Treatment in Subjects With Type 2 Diabetes
Acronym: PREDICTIVE™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1720
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir

SUMMARY:
This trial is conducted in the United States of America (USA). This trial aims for a comparison of the safety and efficacy in subjects with type 2 diabetes using either self titration or physician guided titration according to the local standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes HbA1C <= 12.0% within the past 12 months;
* BMI <= 45.0 kg/m2
* Initiation, addition of, change to, or continuation of basal insulin therapy with insulin detemir as deemed necessary by Investigator

Exclusion Criteria:

* Anticipated change in concomitant medication known to interfere with glucose metabolism such as systemic steroids, non-selective beta-blockers or mono amine oxidase (MAO) inhibitors.
* Proliferative retinopathy or maculopathy that has required acute treatment within the last 6 months.
* Any glucose lowering medication that is not indicated in combination with insulin, such as GLP-1 Analogues
* Known hypoglycemia unawareness or recurrent major hypoglycemia, as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5652 (Actual)
Dates: Start 2005-10; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the change from baseline to end of treatment | after 26 weeks in the value of laboratory-measured HbA1c between the self adjustment versus the standard of care group

SECONDARY OUTCOMES:
Spontaneously reported adverse events during the trial
Incidence of severe hypoglycaemic during the trial nocturnal (11 pm - 6 am)
FPG during the trial (central laboratory) at Visit 2 and Visit 3
Proportion of subjects achieving HbA1C <= 7.0% at Visit 2 and Visit 3
Insulin detemir doses at Visit 2 and Visit 3
Within-subject variation of before-breakfast SMPG values at Visit 2 and Visit 3

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Plainsboro, New Jersey, United States

REFERENCES:
- [Result] Meneghini L, Koenen C, Weng W, Selam JL. The usage of a simplified self-titration dosing guideline (303 Algorithm) for insulin detemir in patients with type 2 diabetes--results of the randomized, controlled PREDICTIVE 303 study. Diabetes Obes Metab. 2007 Nov;9(6):902-13. doi: 10.1111/j.1463-1326.2007.00804.x. PMID 17924873
- [Result] Selam JL, Koenen C, Weng W, Meneghini L. Improving glycemic control with insulin detemir using the 303 Algorithm in insulin naive patients with type 2 diabetes: a subgroup analysis of the US PREDICTIVE 303 study. Curr Med Res Opin. 2008 Jan;24(1):11-20. doi: 10.1185/030079908x242755. PMID 18021495
- [Result] Bhargava A, Chan V, Kimball ES, Oyer DS. Effects of Age on Glycemic Control in Patients With Type 2 Diabetes Treated with Insulin Detemir: A Post-Hoc Analysis of the PREDICTIVE 303 Study. Drugs Aging. 2016 Feb;33(2):135-41. doi: 10.1007/s40266-016-0342-9. PMID 26833348
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com